CLINICAL TRIAL: NCT01444469
Title: A Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy of Oral Azithromycin (500 Mg OD) as a Supplement to Standard Care for Adult Patients With Acute Exacerbations of Asthma
Brief Title: AZithromycin Against pLacebo in Exacerbations of Asthma
Acronym: AZALEA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-001093-26; 10/60/27 (Other Grant/Funding Number: NIHR EME)
Record Dates: First submitted 2011-09-22; First posted 2011-09-30 (Estimated); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Asthma
Keywords: Asthma exacerbations; Respiratory disease; Viral infection; Macrolide/ketolide antibiotics; Mycoplasma pneumoniae (M. pneumoniae); Chlamydophila pneumoniae (C. pneumoniae)
MeSH Terms: conditions — Asthma; Respiration Disorders; Virus Diseases | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithromycin (Zithromax) (Experimental): 500 mg of azithromycin (2×250mg capsules)
  Interventions: Drug: Zithromax
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zithromax — 250mg * 2 capsules once daily for three days
  Other Names: Azithromycin
  Arms: Azithromycin (Zithromax)
Drug: Placebo — Lactose powder
  Arms: Placebo

SUMMARY:
Acute attacks (exacerbations) of asthma are common and cause a great deal of suffering in asthmatic patients. Current treatments for asthma attacks are not completely effective and new and better treatments are needed. Viruses often cause asthma attacks and bacterial lung infections have also been associated with asthma attacks. However, the role for bacteria is uncertain. Current asthma guidelines for doctors treating asthma exacerbations do not recommend the routine use of antibiotics. The investigators would like to investigate whether or not azithromycin, which is a safe and well tolerated antibiotic (an antibacterial) that has been used for many years in the treatment of respiratory disease, might be of benefit in asthma attacks. As there is some evidence that azithromycin has anti-viral properties this may add to its benefits (antibiotics don't usually affect viruses). By looking at the effect of azithromycin on asthma attacks this will help us to show whether or not azithromycin should be recommended during an acute asthma attack in addition to the usual care that is provided to these patients as it may help them recover quicker from the exacerbation. The investigators will also be able to look at why azithromycin may be effective - if it is having an anti-bacterial and/or anti-viral effect.

ELIGIBILITY:
Inclusion criteria

Patients meeting all of the following criteria will be considered for admission to the study:

* Adults, either sex, ages 18-55 years or age 56 to 65 with < 20 pack year smoking history or >65 with <5 pack year smoking history
* Patients with a documented history of asthma for >6 consecutive months, and
* Patients presenting within 48 hours (of initial presentation to medical care) with an acute deterioration in asthma control (increased wheeze, dyspnea and/or cough and/or reduced PEF) and requiring a course of oral steroids
* Patients with a PEF or FEV1 less than 80% of predicted normal or patient's best at presentation, at recruitment or in the time elapsed between presentation and recruitment
* Patients must be able to complete diaries and quality of life questionnaires.
* Patients must sign and date an informed consent prior to any study procedures.

Exclusion criteria

Patients presenting with any of the following will not be included in the study:

* Patients with known prolongation of the QT interval, a history of torsades de pointes, congenital long QT syndrome, bradyarrhythmias or uncompensated heart failure, patients on drugs known to prolong the QT interval and patients with ongoing proarrhythmic conditions such as uncorrected hypokalemia or hypomagnesemia, clinically significant bradycardia, and patients receiving Class IA (quinidine, procainamide) or Class III (dofetilide, aminodarone, sotalol) antiarrhythmic agents.
* Smokers aged 56-65 with a >20 pack year history, or aged >65 with >5 pack year history
* Patients requiring immediate placement in ICU
* Patients who used oral or systemic antibiotics within 28 days prior to enrolment
* Patients with known impaired hepatic function (ALT/AST > 2 ULN)
* Patients with significant lung disease (including COPD) other than asthma
* Patients with > 20mg oral corticosteroid maintenance therapy
* Patients requiring other antibiotic therapy
* Patients who are receiving other medications or who have other disease conditions or infections that could interfere with the evaluation of drug efficacy or safety
* Women who are breast-feeding or are pregnant, as demonstrated by a urine pregnancy test carried out before exposure to study medication or the start of any study procedure that could pose a risk to the foetus
* Patients with suspected or known hypersensitivity to, or suspected serious adverse reaction to Azithromycin or any of the macrolide or ketolide class of antibiotics, erythromycin or to any excipients thereof
* Patients who have received treatment with any other investigational drug within 1 month prior to study entry, or have such treatment planned for the study period during treatment and follow up phase
* Patients with a concomitant condition (including clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic disease) making implementation of the protocol or interpretation of the study results difficult
* Patients with mental conditions rendering them unable to understand the nature, scope, and possible consequences of the study.
* Patients unlikely to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits.
* No subject will be allowed to enrol in this study more than once.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2011-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Diary card summary symptom score | 10 days after randomisation
  Symptoms include wheezing, breathlessness and coughing assessed at 10 days after randomisation.

SECONDARY OUTCOMES:
Quality of life assessed by acute asthma QolQ (Juniper) | 5 & 10 days post randomisation
  * Health status assessed by acute asthma QolQ (Juniper)
  * Health status assessed by Mini Asthma QolQ (Juniper)
Time to 50% reduction in symptom score | From Visit 1 (day 1) to Visit 4 (day 42)
Pulmonary Function tests | 5 & 10 days post randomisation
  Pulmonary function tests include: FEV1, FVC, FEV1/FVC ratio, PEF, FEF25-75% and FEF50%

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian L Johnston, MBBS, PhD, FRCP, Study Chair — Imperial College London
Locations (14):
- United Kingdom (14):
  - Barnsley Hospital NHS Foundation, Barnsley, England
  - Countess of Chester Hospital NHS Foundation Trust, Liverpool, England
  - Surrey & Sussex Healthcare NHS Trust, Redhill, England
  - Heart of England NHS Foundation Trust, Birmingham
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - University of Glasgow, Glasgow
  - University Hospitals of Leicester NHS Foundation Trust, Leicester
  - Imperial College Healthcare NHS Trust, London
  - University Hospital of South Manchester Foundation Trust, Manchester
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - University Hospital of North Tees, Stockton-on-Tees
  - Sherwood Forest Hospitals NHS Foundation Trust, Sutton in Ashfield

REFERENCES:
- [Derived] Johnston SL, Szigeti M, Cross M, Brightling C, Chaudhuri R, Harrison T, Mansur A, Robison L, Sattar Z, Jackson D, Mallia P, Wong E, Corrigan C, Higgins B, Ind P, Singh D, Thomson NC, Ashby D, Chauhan A; AZALEA Trial Team. Azithromycin for Acute Exacerbations of Asthma : The AZALEA Randomized Clinical Trial. JAMA Intern Med. 2016 Nov 1;176(11):1630-1637. doi: 10.1001/jamainternmed.2016.5664. PMID 27653939